CLINICAL TRIAL: NCT03965832
Title: A Pilot Study to Evaluate the Feasibility of Using High-flow Nasal Therapy During Exercise in Patients With Cystic Fibrosis and Severe Lung Disease
Brief Title: HFNT During Exercise in CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RM19/121917; 19/LO/0671 (Other: REC Reference); 262095 (Other: IRAS)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Cystic Fibrosis
Keywords: high-flow nasal therapy; oxygen therapy; Exercise-induced desaturation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNT (Experimental): Patients who meet the eligibility criteria will be randomized to receive HFNT and then crossover to other device during the study procedures.
  Interventions: Device: HFNT during exercise; Device: Standard oxygen therapy/RA
- Standard oxygen (Experimental): Patients who meet the eligibility criteria will be randomized to receive Standard oxygen and then crossover to HFNT during the study procedures.
  Interventions: Device: HFNT during exercise; Device: Standard oxygen therapy/RA

INTERVENTIONS:
Device: HFNT during exercise — 6-minute walking test performed initially on HFNT. HFNT will be set with an inspiratory flow rate at 45-55 L/min (maximal tolerated flow), temperature at 37°C or 34°C if perceived as too warm, and fraction on inspired oxygen (FiO2) as at baseline conditions during exercise.
  Participants will then cross-over to repeat the test on baseline conditions.
Device: Standard oxygen therapy/RA — 6-minute walking test performed on baseline conditions. Participants will then be cross over to repeat the test on HFNT

SUMMARY:
Cystic fibrosis (CF) is a genetic condition characterised by recurrent lung infections, inflammation and progressive lung damage. Patients with CF and advanced lung disease are limited when exercising and performing activities of daily life, due to increased breathlessness and lower oxygen levels.

Exercise is an important part of treatment in CF, having been shown to slow down the lung disease and improve quality of life. Patients with CF are encouraged to exercise both at home and during hospital admissions, even when the lung disease is advanced. Often, oxygen therapy is used in patients whose oxygen levels are otherwise too low during. This, however, does not improve their breathlessness.

Recently, a device to deliver air at flows higher than what other device allow has become available. High flow nasal therapy (HFNT) provides patients with air or a blend of air and oxygen at flows up to 60 L/min. HFNT can improve oxygen levels and reduce shortness of breath in many situations both in the acute and chronic setting. HFNT was shown to improve the tolerance to exercise in patients with other respiratory conditions (chronic obstructive pulmonary disease).

In CF, HFNT is routinely used for patients admitted with acute respiratory failure (inability to maintain adequate oxygenation) with positive results.

In this study, the Investigators aim to understand if HFNT can improve the exercise tolerance in patients with CF and advanced lung disease, by reducing breathlessness and avoiding the drop in oxygenation observed during simple training.

The Investigators propose a short study to assess if further large clinical trials are feasible and practical, and will therefore collect preliminary data to have some results to use for planning other studies. All patients who are admitted in the Leeds Regional Adult CF Unit will be considered for participation in the study.

DETAILED DESCRIPTION:
Regular high-level exercise in people with CF has been linked with reduced rate of decline in lung function, is positively related to quality of life and improvement in bone mineralisation. Unfortunately, exercise tolerance in patients with cystic fibrosis (CF) and severe lung disease is limited by dyspnoea, exercise-induced desaturations (EID) and fatigue. Therefore, a reduction in patients' activity level can be observed, which would lead to further deconditioning.

High-flow nasal therapy (HFNT) delivers heated, humidified and oxygenated gas with flow rates up to 60 L/min at FIO2 adjustable between 0.21 and 1.0 via soft, loose fitting, large bore nasal prongs (Airvo2/OptiflowTM). HFNT has been shown to (a.) Wash out nasopharyngeal dead space, minimizing rebreathing of CO2 and acting as a reservoir for fresh air, thus contributing to improved gas exchange with respect to CO2 and O2. (b) Lower respiratory rate and provide a small positive end expiratory effect. (c) Provide oxygenated gas at a flow that matches more closely the patient's spontaneous inspiratory flow rate, thus attenuating inspiratory resistance within the nasopharynx and eliminating the related increase in work of breathing. (d) Provide warmed and humidified gas (37°C and 44 mg/L H2O) thus reducing airway dryness, enhancing patient comfort and reducing the metabolic work associated with gas conditioning. (e) Moisten secretion and facilitate mucociliary clearance.

HFNT is being extensively studied, in comparison to NIV and conventional oxygen therapy, in de novo acute respiratory failure, in post-surgical and post-extubation setting and in do-not-intubate patients. One pilot study has demonstrated that HFNT can increase exercise tolerance in stable patients with severe COPD, with improvement in oxygen saturation and perceived dyspnea and muscle fatigue.

As the main limiting factors for exercise tolerance in patients with CF and severe lung disease are perceived dyspnoea, and hypoxaemia related symptoms, secondary to static and dynamic hyperinflation, it is conceivable that HFNT could have beneficial effects in improving exercise tolerance and reducing symptoms.

The Investigators propose here a pilot study to assess a feasibility of a subsequent trial of long-term use of HFNT during exercise training in patients with CF compared to standard oxygen or room air.

A single-centre, short-term, open, randomized, cross-over study is planned. The Investigators will compare the results of 6-MWT on HFNT and without HFNT (either on conventional oxygen therapy or room air). The Investigators plan to enroll 25 subjects, expecting a drop-out rate of 5%, to have 20 subjects completing the study. Each subject will serve as their own control.

Participants in the study will be asked to fill in a questionnaire which is routinely used in the assessment of exercise and activity among patients with CF, and has been previously validated in other CF Centre.

Study procedures will consist in:

* Two 6-minute walking test (24 to 48 hours apart). The 6-minute walking test is a simple assessment of exercise and consist in the patient having a brisk walk for 6 minutes. Patients can increase or decrease the speed at their will while walking. Oxygen and carbon dioxide (the waste gas) levels will be measured through a sensor applied to the skin. Patients will be asked to score their breathlessness, comfort and fatigue, before, during and after the test. One of the tests will be performed under the usual condition, the other test on HFNT.
* Lung function before and after each 6-minute walking test. Lung function is a standard assessment in CF, consisting in blowing air into a machine to measure lung volumes and flows.

Measures related to the 6-minute walking test and the lung function will be recorded as part of the study. The Investigators will record patients' feedback on shortness of breath, comfort and fatigue, but also oxygen and carbon dioxide levels, frequency of breathing and distance walked during the 6 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF
* Severe lung disease (FEV1 ≤40%)

Exclusion Criteria:

* Acute viral illness
* Requirements of >6 L/min nasal O2 to maintain SpO2 >88% at rest
* Acute respiratory acidosis
* Arthritis exacerbation
* Inability to obtain informed consent
* Recent pneumothorax (<6 weeks)
* Usual contraindication to exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
6 minute walking distance | 6 minutes
  Change in the 6 minute walking distance (exploratory outcome of interest)

OTHER OUTCOMES:
Oxygen saturation (SpO2) | 6 minutes
  Mean and Nadir SpO2 during 6MWT (exploratory outcome of interest)
Time to recovery - SpO2 | 30 minutes
  Time to recovery for SpO2 at end of exercise (exploratory outcome of interest)
Transcutaneous CO2 | 6 minutes and during recovery time (30 minutes)
  Mean tCO2 (exploratory outcome of interest)
Respiratory rate (RR) | 6 minutes and during recovery time (10 minutes)
  (exploratory outcome of interest)
Dyspnea | 6 minutes and during recovery time (10 minutes)
  Measured with Borg score (exploratory outcome of interest): 0 no breathlessness to 10 maximal breathlessness
Fatigue | 6 minutes and during recovery time (10 minutes)
  Measured with Borg score (exploratory outcome of interest): 0 no fatigue at all to 10 maximal fatigue
Comfort | 6 minutes and during recovery time (10 minutes)
  Measured with VAS (exploratory outcome of interest): 0 most uncomfortable to 10 very comfortable

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Spoletini, Principal Investigator — LTHT; Daniel G Peckham, Principal Investigator — LTHT
Locations (1):
- St James's University Hospital, Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Background] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Background] Sklar MC, Dres M, Rittayamai N, West B, Grieco DL, Telias I, Junhasavasdikul D, Rauseo M, Pham T, Madotto F, Campbell C, Tullis E, Brochard L. High-flow nasal oxygen versus noninvasive ventilation in adult patients with cystic fibrosis: a randomized crossover physiological study. Ann Intensive Care. 2018 Sep 5;8(1):85. doi: 10.1186/s13613-018-0432-4. PMID 30187270
- [Background] Cirio S, Piran M, Vitacca M, Piaggi G, Ceriana P, Prazzoli M, Paneroni M, Carlucci A. Effects of heated and humidified high flow gases during high-intensity constant-load exercise on severe COPD patients with ventilatory limitation. Respir Med. 2016 Sep;118:128-132. doi: 10.1016/j.rmed.2016.08.004. Epub 2016 Aug 8. PMID 27578482
- [Derived] Spoletini G, Watson R, Lim WY, Pollard K, Etherington C, Clifton IJ, Peckham DG. Nasal high-flow therapy as an adjunct to exercise in patients with cystic fibrosis: A pilot feasibility trial. J Cyst Fibros. 2021 Sep;20(5):e46-e52. doi: 10.1016/j.jcf.2021.03.005. Epub 2021 Apr 1. PMID 33814320